CLINICAL TRIAL: NCT01147354
Title: Effect of Selenium Supplementation on Inflammatory,Oxidative and Nutritional Markers in Hemodialysis Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zahra Sohrabi (Other)
Collaborators: Shiraz University of Medical Sciences (Other)
Responsible Party: Sponsor-Investigator, Zahra Sohrabi, Ph.D, Shiraz University of Medical Sciences
Organization: Shiraz University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 88-4747
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Inflammation; Malnutrition; Complication of Hemodialysis
Keywords: Hemodialysis; oxidative stress; selenium; inflammation
MeSH Terms: conditions — Inflammation; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group (Experimental): The patients in this arm took 200 micrograms of selenium yeast daily for 12 weeks.
  Interventions: Dietary Supplement: selenium yeast
- control group (Placebo Comparator): The patients in this arm took one placebo capsule daily for 12 weeks.
  Interventions: Other: placebo capsules

INTERVENTIONS:
Dietary Supplement: selenium yeast — The patients in this arm took 200 micrograms of selenium yeast daily for 12 weeks.
  Arms: experimental group
Other: placebo capsules — The patients in this arm took one placebo capsule daily for 12 weeks.
  Arms: control group

SUMMARY:
The aim of this study is to evaluate the effect of selenium supplementation on oxidative, inflammatory and nutritional markers in hemodialysis patients.

DETAILED DESCRIPTION:
After screening all of 280 patients under regular HD in Faghihi Hospital Hemodialysis Center, 80 stable patients in the age range of 18-80 years old were found to be eligible for enrollment and gave their informed consent to participate in this trial. Subjects were excluded if they were prescribed any multivitamins or immunosuppressive drugs or taking antioxidant supplements including vitamin E, vitamin C, lipoic acid, omega-3 fatty acids, soy extracts and green-tea preparations within 2 months prior to enrollment in the study or if they had been hospitalized in the previous month, we also excluded the ones who were pregnant or had active infections. The Ethics Committee of Shiraz University of Medical Sciences reviewed and approved the protocol of this study.These patients were randomly assigned in a 1:1 ratio into 2 groups of selenium(200µg) or placebo and were followed for 12 weeks.In order to determine the nutritional statuses of all patients, at the baseline, the questions of SGA and MIS questionnaire were read to the patients and completed in person by the main investigator. The questions of SGA and MIS were also asked by the same person at the end of treatment phase.Before the onset of the treatment and after the end of the treatment phase of the study, 10cc blood samples were taken from each patient.The blood was taken from the patient's arm used for hemodialysis cannula just before the beginning of the hemodialysis procedure. The serum was separated by centrifugation at 3000 g/min for 5 min and stored at -70°C. Serum levels of malondialdehyde (MDA), interleukin-6 (IL-6), high sensitive C-reactive protein (HSCRP), ferritin, transferrin, homocysteine, calcium , phosphate, parathyroid hormone (PTH), albumin, blood urea nitrogen (BUN), and creatinine as well as hemoglobin (Hb) levels were measured in all patients at the baseline and at the end of treatment phase of study.The aim of this study was to evaluate the effect of selenium supplementation on oxidative, inflammatory and nutritional markers in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were dialyzed three times a week at least for 3 months or more

Exclusion Criteria:

* Patients who took any multivitamins or immunosuppressive drugs within 2 months prior to enrollment in the study
* Patients consuming antioxidant supplements including vitamin E, vitamin C, lipoic acid,omega-3 fatty acids, soy extracts and green-tea preparations within 2 months prior to enrollment in the study
* Patients who were Hospitalized in the previous month
* Patients who had active infections
* Being pregnant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Subjective Global Assessment | 12-weeks
  changes in nutritional status according to SGA from baseline to end of treatment

SECONDARY OUTCOMES:
serum albumin | 12-weeks
hemoglobin | 12-weeks
serum malondialdehyde | 12-weeks
serum parathyroid hormone | 12-weeks
serum interleukin-6 | 12-weeks
serum phosphorus | 12-weeks
serum high sensitive c-reactive protein | 12-weeks
serum calcium | 12-weeks
serum lipoproteins | 12-weeks
serum ferritin | 12-weeks
serum homocysteine | 12-weeks
total iron binding capacity (TIBC) | 12-weeks
body mass index (BMI) | 12-weeks
malnutrition-inflammation score (MIS) | 12-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Sohrabi, Ph.D, Principal Investigator — Shiraz University of Medical Sciences; Mohammad mahdi Sagheb, M.D, Study Chair — Shiraz University of Medical Sciences; Moosa Salehi, Ph.D, Principal Investigator — Shiraz University of Medical Sciences; Maryam Ekramzadeh, Ph.D, Principal Investigator — Shiraz University of Medical Sciences; Mohammad Kazem Fallahzadeh, M.D, Principal Investigator — Shiraz University of Medical Sciences; Maryam Ayatollahi, Ph.D, Principal Investigator — Shiraz University of Medical Sciences; Bita Geramizadeh, M.D, Principal Investigator — Shiraz University of Medical Sciences; Jafar Hassanzadeh, Ph.D, Principal Investigator — Shiraz University of Medical Sciences
Locations (1):
- Shiraz University of Medical Sciences, Shiraz, Fars, Iran

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745